CLINICAL TRIAL: NCT06870643
Title: Effect of Parabiotics As an Adjuvant in Nutritional Management of Pediatric Celiac Patients
Brief Title: Parabiotics Use with Nutritional Management in Pediatric Celiac Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Haya Essam Ibrahim, lecturer of pediatrics, Ain Shams University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: FMASU M S 697/2022
Record Dates: First submitted 2025-03-06; First posted 2025-03-11 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Celiac Disease in Children
MeSH Terms: interventions — Diet, Gluten-Free

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pediatric celiac patients (Experimental): Strict gluten free food regimen for 3 weeks then parabiotics (Lacteolfort ®) added for another 3 weeks.
  Interventions: Other: Gluten free diet for 3 weeks then parabiotic (Lacteolfort®) for another 3 weeks

INTERVENTIONS:
Other: Gluten free diet for 3 weeks then parabiotic (Lacteolfort®) for another 3 weeks — Gluten free diet for 3 weeks then parabiotic (Lacteolfort®) for another 3 weeks.

SUMMARY:
This is a sequential study to evaluate the effect of parabiotics as an adjuvant therapy with gluten restriction on quality of life in children with Celiac disease.

ELIGIBILITY:
Inclusion Criteria:

• Celiac cases diagnosed either by non-biopsy approach {serology based: high IgA antibodies against transglutaminase ≥10 times the upper limit of normal with positive endomysial antibodies or diagnosed by biopsy using March classification

Exclusion Criteria:

* Immunocompromised patients
* Patients taking immunosuppressant drugs or antibiotics within the last 4 weeks or during the study

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2023-07-12 (Actual); Primary Completion 2024-12-26 (Actual); Study Completion 2025-02-20 (Actual)

PRIMARY OUTCOMES:
Evaluate the effect of parabiotics as an adjuvant on celiac patients' quality of life . | 3 weeks
  Evaluate the effect of parabiotics as an adjuvant therapy to gluten free diet in celiac patients' quality of life using pediatric quality of life(PedsQL)Gastrointestinal symptoms module version 3.0. It has specific gastrointestinal symptom domains, scoring from 0-4 (0 indicates never a problem, 1 indicates almost never a problem, 2 indicates sometimes a problem, 3 indicates often a problem and 4 indicates almost always a problem) then cores are transformed on a scale from 0 to 100. Items are reverse scored and linearly transformed to a 0-100 scale as follows: 0=100, 1=75, 2=50, 3=25, 4=0. The higher the score is the better quality of life, there is no cutoff value for this score.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Abbassia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided